CLINICAL TRIAL: NCT06633926
Title: Integrative Approaches for Cancer Survivorship: A Multi-Site Feasibility and Acceptability Study (Aim 2)
Brief Title: Integrative Approaches for Cancer Survivorship (IACS3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24807; NCI-2024-07529 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP)); R01AT012522 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
Keywords: Health Intervention
MeSH Terms: interventions — Nutrition Assessment; Yoga; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to the study hypothesis. Research staff involved with data analysis will be blinded to group assignment until the database is locked. The statistician will remain blinded until the completion of the analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ayurveda and Usual Care (AVI) (Experimental): Participants receive usual care on study. Participants also receive nutrition education, lifestyle recommendations, and participate in yoga, as well as marma therapeutic touch during one-on-one AVI visits over 1-2 hours for up to 14 visits over 6 months. After 6 months, participants may also complete a videoconference visit over 30 minutes once monthly for 6 months. In addition, participants will complete online questionnaires at baseline and at the end of 6 months.
  Interventions: Behavioral: Nutrition Education; Behavioral: Lifestyle Counseling; Other: Yoga; Procedure: Marma therapy; Other: Quality of Life Questionnaire Administration
- Health Education and Usual Care (HEI) (Experimental): Participants receive usual care on study. Participants also attend online HEI sessions over 1 hour each for up to 15 sessions over 6 months. In addition, participants will complete online questionnaires at baseline and at the end of 6 months.
  Interventions: Other: Educational Intervention; Other: Quality of Life Questionnaire Administration

INTERVENTIONS:
Behavioral: Nutrition Education — Given nutrition education
  Arms: Ayurveda and Usual Care (AVI)
Behavioral: Lifestyle Counseling — Given lifestyle recommendations
  Arms: Ayurveda and Usual Care (AVI)
Other: Yoga — Participate in yoga
  Other Names: Yoga therapy
  Arms: Ayurveda and Usual Care (AVI)
Procedure: Marma therapy — Participate in marma therapeutic touch
  Other Names: Marma therapeutic touch therapy; Therapeutic touch therapy
  Arms: Ayurveda and Usual Care (AVI)
Other: Educational Intervention — Attend online HEI sessions
  Other Names: Education for Intervention
  Arms: Health Education and Usual Care (HEI)
Other: Quality of Life Questionnaire Administration — Self-reported questionnaires are given to participants to complete
  Other Names: Quality of Life Survey

SUMMARY:
This clinical trial is a two-arm pilot randomized controlled trial for non-metastatic breast cancer survivors to determine the feasibility, acceptability, and fidelity of two integrative health approaches and study design in a multi-site setting. Participants (n=104) will be randomized to either the Ayurveda Intervention (AVI) or Facing Forward Health Education Intervention (FFHEI). Integrative health combines biomedical and complementary approaches together in a coordinated way. AVI, a multi-modal intervention, includes nutritional education, lifestyle practices, yoga, and therapeutic touch, called marma, to help the body and mind feel balanced. FFHEI provides health education using self-directed online content and interactive videos based on the latest science in cancer survivorship. This study does not intend to conduct tests of efficacy and is focused on feasibility outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

I. Determine feasibility and acceptability of this design in a multi-site setting.

SECONDARY OBJECTIVES

I. Evaluate Quality of Life (QOL).

II. Evaluate Cancer Associated Symptoms.

OUTLINE: Participants are randomized in a 1:1 ratio to 1 of 2 arms.

ARM I: Participants receive usual care on study. Participants also receive nutrition education, lifestyle recommendations, and participate in yoga, as well as marma therapeutic touch during one-on-one AVI visits over 1-2 hours for up to 14 visits over 6 months. After 6 months, participants may also complete a videoconference visit over 30 minutes once monthly for 6 months.

ARM II: Participants receive usual care on study. Participants also access self-directed online HEI sessions over 1 hour each for up to 15 sessions over 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Able to read, write, and understand English.
4. Ability of individual or legal guardian/representative to understand a verbal informed consent document, and the willingness to sign it.
5. Non-metastatic breast cancer patients who are between 1 and 36 months after completion of primary treatment (i.e., surgery, radiotherapy, chemotherapy) and are in a complete remission.
6. Participants should have received chemotherapy as part of their primary treatment.
7. Have an impaired quality of life (report a score of 5 or less on question 30 of the European Organisation for Research and Treatment of Cancer Quality of Life Cancer questionnaire (EORTC-QLQ-C30). "How would you rate your overall quality of life during the past week?"
8. Karnofsky Performance Status Score (KPS) >=60

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.
2. Metastatic disease and receiving chemotherapy or radiotherapy at the time of study enrollment (participants with non-metastatic disease who are receiving anti-Her2 directed treatment alone in the adjuvant setting are eligible).
3. Participants are within 1 month after surgery for cancer, including breast reconstructive surgery but not including implant exchange.
4. Cancer surgery planned during the initial 6-month study period.
5. Been on adjuvant hormone therapy (for breast cancer) less than 2 months at the time of enrollment.
6. Received Ayurvedic treatment during the 3 months preceding enrollment.
7. If a participant reports severe anxiety or depression, has severe depression assessed by Patient Health Questionnaire (PHQ)-9 using a cut-off of 20 or higher, or severe anxiety assessed by the General Anxiety Disorder-7 (GAD-7) using a cut-off 15 or higher.
8. Current suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of all screened participants who were ultimately enrolled | Up to 15 months
  The proportion of all screened participants who were ultimately enrolled onto the study will be reported.
Proportion of eligible screens who decline to enroll | Up to 15 months
  Proportion of eligible screens who decline to enroll due to concerns about randomization will be reported.
Proportion of enrolled participants who drop out immediately after assignment | Up to 15 months
  Proportion of enrolled participants who drop out after learning their randomization assignment will be reported.
Proportion of randomized participants who drop out during participation | Up to 6 months
  Proportion of randomized participants who drop out after participating in the study interventions due to unhappiness with randomization assignment will be reported.
Retention rates | Up to 6 months
  The proportion of participants who complete <=70% of study measures will be reported.
Adherence to intervention rate | Up to 6 months
  Proportion of participants who attended at least 10 out of 14 sessions or completed 10 out of 14 HEI sessions (≥80%) will be reported
Practitioner fidelity rates | Up to 6 months
  Fidelity of adherence to the intervention will be assessed through a contact check-list method comparing the intervention to the study manuals and the rate of adherence will be reported.
Assessment completion rates | Up to 6 months
  Assessment completion rates will be defined as the percentage of participants completing each assessment.
Mean scores on an Acceptability of Intervention measure | Up to 6 months
  The measure used for this study is a single item assessment of the implementation to participants perceived acceptability of the intervention. The response item response falls on a numeric rating scale of 0 to 10. A mean score is calculated by averaging responses from all participants. The intervention will be determined acceptable if the overall mean score is >= 8.
Change in mean scores on an Expectation of Benefit questionnaire over time | Up to 6 months
  The change in participant's expectation of intervention benefit at baseline-pre and post randomization-will be assessed using a 0-10 numeric rating scale of 0 to 10. A mean score is calculated by averaging responses from all participants. The instrument for expectancy, is adapted from a measure created by Kalauokalani et. al, with higher scores indicating a higher level of expectation that the intervention will be beneficial.

SECONDARY OUTCOMES:
Mean scores on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-C30)-Functional Domains over time | Up to 6 months
  The functional domains measure the quality of life in Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning. Scores consists of responses to items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning
Mean scores on the EORTC-C30 Global Health Status scale over time | Up to 6 months
  The global health status score consists of responses to two items with responses ranging from 1="very poor" to 4="excellent". The raw score is calculated by estimating the mean of the two items that make up the global health scale with a resulting total range of 1-7. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the global health status represents a higher quality of life.
Mean scores on the EORTC-C30 Breast Cancer (BR42) subscales scale over time | Up to 6 months
  The breast cancer module of the EORTC-C30 (BR42) status score consists of responses to 42 items divided into 10 scales: Breast Symptoms, Body Image, Sexual Functioning, Arm Symptoms, Systemic Chemotherapy Side Effects, Hand/Feet Symptoms/Neuropathy, Skeletal Symptoms, Endocrine Symptoms, Breast Satisfaction, Vaginal Symptoms, and 3 single items: Weight Gain, Sexual Enjoyment and Future Perspective with responses ranging from 1="very poor" to 4="excellent". The raw score is calculated by estimating the mean of the items that make up the scales with a resulting total range of 1-168. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score represents a higher quality of life.
Mean scores on the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue scale over time | Up to 6 months
  This 6-item questionnaire to measure fatigue based on responses to statements about how the participants feel with a response ranging from 1="Never" to 5="Always", and a total raw score ranging from 6 - 30, which are converted to a scaled T-score (range 33.4 to 76.8) with higher scores indicating a greater feeling of fatigue.
Mean scores on the PROMIS Sleep Disturbance scale over time | Up to 6 months
  This 6-item questionnaire to measure sleep disturbance based on responses to statements about how the participants feel with a response ranging from 1="Never" to 5="Always", and a total raw score ranging from 6 - 30, which are converted to a scaled T-score (range 31.7 to 73.3) with higher scores indicating a greater feeling of sleep disturbance.
Mean scores on the PROMIS Anxiety scale (Short Form) over time | Up to 6 months
  The PROMIS Anxiety Short form consists of 2 items addressing patient anxiety with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of anxiety.
Mean scores on the PROMIS Depressive symptoms scale over time | Up to 6 months
  The PROMIS Depression Short form consists of 4 items addressing patient depression with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of depression.
Mean scores on the PROMIS Pain scale over time | Up to 6 months
  This 4-item questionnaire to measure the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities based on responses to statements about how the participants feel with a with a response ranging from 1="Never" to 5="Always", and a total raw score ranging from 4 - 20, which are converted to a scaled T-score (range 41.6 to 75.6) with higher scores indicating a greater hinderance to engagement in activities based on how much pain participants are experiencing.
Mean scores on the PROMIS Self Efficacy over time | Up to 6 months
  This 4-item questionnaire to measure the extent to which persons with chronic conditions are able to managing daily activities, medications and treatments, symptoms, emotions, and social interactions based on responses to statements about how the participants feel with a with a response ranging from 1="I am not at all confident" to 5="I am very confident", and a total raw score ranging from 4 - 20, which are then converted to a scaled T-score (range 18.6 to 64.7) with higher scores indicating a greater feeling of self-efficacy in managing daily activities.
Mean scores on the Functional Assessment of Chronic Illness Therapy- Spiritual Well-Being measure (FACIT-SP-12) over time | Up to 6 months
  The FACIT-SP-12 is a 12-item questionnaire which measures a participant's spiritual well-being for the past 7 days. Item responses range from 0 (not at all) to 4 (very much). The sum of item scores is used to calculate a total FACIT-SP-12 score ranging from 0 to 48. The higher the score, the better the QOL/spiritual well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Dhruva, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - Zuckerberg San Francisco General, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Kaiser Permanente Northwest (KPNW), San Francisco, California
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared with research collaborators
Supporting Information: Study Protocol, SAP